CLINICAL TRIAL: NCT05181995
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of 50 mg NYX-783 Once Daily Compared to Placebo in Participants With Post-Traumatic Stress Disorder (PTSD)
Brief Title: Safety and Efficacy of 50 mg NYX-783 QD vs. Placebo in PTSD
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: company decision
Sponsor: Aptinyx (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NYX-783-2009
Record Dates: First submitted 2021-12-15; First posted 2022-01-10 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 50 mg NYX-783 QD (Experimental): 50 mg NYX-783 QD
  Interventions: Drug: NYX-783
- Placebo (Placebo Comparator): Placebo QD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NYX-783 — NYX-783
  Arms: 50 mg NYX-783 QD
Drug: Placebo — Placebo for 50 mg NYX-783
  Arms: Placebo

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of 50 mg NYX-783 Once Daily Compared to Placebo in Participants with Post-Traumatic Stress Disorder (PTSD)

ELIGIBILITY:
Inclusion Criteria:

* PTSD (DSM-5 criteria)
* Stable allowed medications with no planned changes from 30 days prior to screening through study participation
* Willing to use highly effective birth control
* Willing to comply with protocol visits and procedures

Exclusion Criteria:

* Moderate to severe traumatic brain injury
* Other psychiatric disorders (based on SCID-5-CT) or neurodegenerative disorders
* Substance use disorder or alcohol use disorder within 6 months prior to screening
* Psychotherapy or cognitive based therapy within 30 days prior to screening
* Use of investigational drug within 30 days prior to screening
* Prior participation in study of NYX-783, NYX-2925 or NYX-458.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
CAPS-5 (Clinician-Administered PTSD Scale for the Diagnostic and Statistical Manual of' Mental Disorders, 5th edition) | study endpoint, up to 10 weeks
  Change from Baseline in CAPS-5

SECONDARY OUTCOMES:
CGI-S (Clinician Global Impression - Severity) | study endpoint, up to 10 weeks
  Change from Baseline in CGI-S
PGI-S (Patient Global Impression - Severity) | study endpoint, up to 10 weeks
  Change from Baseline in PGI-S
SDS (Sheehan Disability Scale) | study endpoint, up to 10 weeks
  Change from Baseline in SDS

CONTACTS AND LOCATIONS:
Locations (36):
- United States (36):
  - Aptinyx Clinical Site, Tuscaloosa, Alabama
  - Aptinyx Clinical Site, Phoenix, Arizona
  - Aptinyx Clinical Site, Bentonville, Arkansas
  - Aptinyx Clinical Site, Bellflower, California
  - Aptinyx Clinical Site, Glendale, California
  - Aptinyx Clinical Site, La Jolla, California
  - Aptinyx Clinical Site, Oceanside, California
  - Aptinyx Clinical Site, Riverside, California
  - Aptinyx Clinical Site, Santa Ana, California
  - Aptinyx Clinical Site, Temecula, California
  - Aptinyx Clinical Site, Torrance, California
  - Aptinyx Clinical Site, Colorado Springs, Colorado
  - Aptinyx Clinical Site, Denver, Colorado
  - Aptinyx Clinical Site, Hialeah, Florida
  - Aptinyx Clinical Site, Hollywood, Florida
  - Aptinyx Clinical Site, Jacksonville, Florida
  - Aptinyx Clinical Site, Jupiter, Florida
  - Aptinyx Clinical Site, Miami, Florida
  - Aptinyx Clinical Site, Miami Lakes, Florida
  - Aptinyx Clinical Site, Okeechobee, Florida
  - Aptinyx Clinical Site, Orlando, Florida
  - Aptinyx Clinical Site, Atlanta, Georgia
  - Aptinyx Clinical Site, Boston, Massachusetts
  - Aptinyx Clinical Site, Las Vegas, Nevada
  - Aptinyx Clinical Site, Albuquerque, New Mexico
  - Aptinyx Clinical Site, New York, New York
  - Aptinyx Clinical Site, Cincinnati, Ohio
  - Aptinyx Clinical Site, Dayton, Ohio
  - Aptinyx Clinical Site, Kettering, Ohio
  - Aptinyx Clinical Site, North Canton, Ohio
  - Aptinyx Clinical Site, Media, Pennsylvania
  - Aptinyx Clinical Site, Memphis, Tennessee
  - Aptinyx Clinical Site, Austin, Texas
  - Aptinyx Clinical Site, Fort Worth, Texas
  - Aptinyx Clinical Site, Houston, Texas
  - Aptinyx Clinical Site, Plano, Texas

IPD SHARING:
Plan to Share IPD: No